CLINICAL TRIAL: NCT05014854
Title: Effects, Acceptance and Usability of a Pressuresensitive Pen and Its Tablet-app in Children With Problematic Fine and Graphomotor Function, Their Occupational Therapists and Their Guardians
Brief Title: SensoGrip - a Pressuresensitive Writing System
Acronym: SensoGrip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FH Campus Wien, University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Othmar Schuhfried, External Lecturer, FH Campus Wien, University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK_21_042_0321
Record Dates: First submitted 2021-08-03; First posted 2021-08-20 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Developmental Delay in Fine Motor Function (Disorder)
Keywords: Occupational Therapy; Handwriting; Children; Writing Pressure; Graphomotor Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Finger and tip pressures are assessed in two phases (A/B). Baseline measurements (A) are collected in the 1st and 2nd therapy session after inclusion. First, data is collected via SEMS (from 2nd grade) or via a sheet with standard forms (1st grade), followed by the recording of a standard sentence (from SEMS) or a standard form at the end of the session. The 2nd session is started and ended with the writing of the chosen standard set. Phase-A-measurements are recorded without feedback.
  From the 3rd therapy session on SensoGrip is used with activated feedback (B). At the end of each session, the same standard set used in Phase A is written twice - once with and once without feedback. This order changes each time to minimize possible bias due to habitation to writing with SensoGrip. Data is recorded in both forms. Children can take SensoGrip home from the 4th session on and use it in daily life.
  In the last session, SEMS or the standard forms are re-executed as initially applied.
  Interventions: Device: Usage of the SensoGrip-System comprised of the SensoGrip pen and a tablet app.

INTERVENTIONS:
Device: Usage of the SensoGrip-System comprised of the SensoGrip pen and a tablet app. — Intervention consists of the usage of the SensoGrip-System in at least 6 and up to 8 therapy session together with the participating child. It is assumed that the standard frequency of therapy sessions is once a week, resuming in a span of 6-8 weeks. 10 minutes of every therapy session during the intervention phase must involve the application of the SensoGrip-System. Sample exercises are made available, therapists can freely choose which exercises are used.

SUMMARY:
The presented study deals with the technically supported, fine motor adjustment of finger and tip pressure in children with graphomotor difficulties by means of a pressure-sensitive pen and a corresponding tablet app. Three target groups (occupational therapists, children, and legal guardians, n=15 each) will be recruited and included in a mixed-methods study. The guiding research questions deal with the effects, acceptance and usability of the applied system.

The active phase of the study covers a period of three months. Expected results lie primarily in the area of improving the target group writing skills (children) and improving opportunities in occupational therapy.

DETAILED DESCRIPTION:
Background

The development of writing competence is not only important for strengthening a child's self-confidence, but is also seen as an essential cornerstone for scholastic (Sassoon, 1990; Stewart, 1992) and academic (Kruse, 1999) success.

A 2015 survey conducted in Germany involving 2000 teachers working in elementary and secondary schools showed that more than 60% of the children are unable to write persistently (Diaz Mayer et al., 2017). As main causes teachers cited hand spasms (73%) and incorrect pen posture (68%). In a longitudinal study in Norway, it was found that 27% of first grade children have problems with handwriting (Karlsdottir & Stefansson, 2002). In the United States and Canada, handwriting problems are one of the most common reasons for referral to school-based occupational therapy (Hoy et al., 2011; Schneck & Case- Smith, 2015). In a survey conducted in Austria, 73% of the occupational therapists indicated that children with circumscribed developmental coordination disorder (DCD) with a referral diagnosis of "problems in fine and/or graphomotor skills" receive occupational therapy (Dolezal & Schönthaler, 2018). Internationally, the prevalence of children with DCD is thought to range from 2% to 20% (Blank & Vinçon, 2020), of which the most common emerging range in literature is 5% - 6% (Gaines et al., 2008; Blank et al., 2012; American Psychiatric Association, 2013).

The perceptual-motor ability of handwriting is based on a complex processing construct that includes inputs from visual-motor coordinative skills, motor planning, cognitive and perceptual abilities, as well as tactile and kinesthetic perceptions (Maeland,1992). Handwriting thus requires very fine motor skills; an exact dosage of the finger pressure on the pencil and the mine pressure on the paper are essential components of writing. The objective of acquiring writing skills is to produce legible, fluent, low-fatigue, efficient, and individualized handwriting (Diaz Mayer et al, 2017). Lin et al (2017) observed that children exhibit difficulty in dosage of applied pressure. Hence, in order to carry out appropriate interventions to improve motor control, it is necessary to collect and integrate all data relevant to pressure. Currently, there is no occupational therapy tool that measures pressure at the pencil tip and at the holding surface. The aim of this project is the interdisciplinary development of a pressure-sensitive pen and associated tablet app as a contribution to digitalization in healthcare. Both parts of the system are the subject of the study, are accordingly in further development and are not commercially available.

Description of the technology used

The system does not ask for personal data and intends to support children who have difficulties in pressure dosage to improve their graphic motor skills through feedback. The procedure is as follows:

* The settings of the pen (pressure range, feedback options: Color, feedback behavior) can be configured and changed via the app.
* Pressure sensors in the pen and on the grip surface of the pen measure the strength of the pressure and the finger pressure.
* Collected data is transferred to the app, displayed and saved.
* Based on the undertaken pen settings, feedback is given via a feedback feature attached to the pen tip (depending on the pressure, the illumination of a ring behind the pen tip varies) in case of individually appropriate pressure conditions.
* Pressure histories recorded during writing are made available for therapeutic decision making via the tablet app.

Study Overview

In order to obtain information about the user experience and user acceptance as well as the effects of the developed system, a mixed-methods approach is followed in this study.

An initial participatory design and development process based on the relevant user groups (occupational therapists, children) and an evaluation process based on all user groups (occupational therapists, children, legal guardians) ensure the usability and acceptance of the project outcome.

Quantitative data will be generated by measuring the pressure data during the writing process. In addition, acceptance factors are quantitatively collected by means of questionnaires based on the "Usefulness, Satisfaction, and Ease of Use Questionnaire" (USE) and the "Unified Theory of Acceptance and Use of Technology 2" (UTAUT2). While the study duration is three months, writing data per participating child will be collected over a duration of eight therapy sessions, usually within eight weeks, due to a rolling recruitment procedure. At the beginning of the intervention phase, the pen and mine pressures of each participating child will be collected as a baseline, without activation of the feedback system integrated in the pen, at four time points each. For this purpose, a sheet with standard forms is used for the first measurement point for children in the 1st grade. For children in the 2nd grade and above, the test procedure "Systematic Assessment of Motor Writing Disorders" (SEMS) is applied. For the later measuring time points a standard sentence from the SEMS is used. The quantitative writing data collected within the regular occupational therapy sessions consist - depending on the school level - of the collection of standard forms or a standard sentence, which are recorded at the beginning and end of the therapy session with and without pen feedback. Familiarity with the system is ensured by means of a minimum duration of use of the SensoGrip-System (10 minutes per session). Qualitative information will be obtained and evaluated via interviews and focus groups with occupational therapists and children after the intervention phase.

Study objectives and research questions

The study aims to achieve the following effects:

* Feedback of the pen supports the child to acquire better graphomotor skills
* The system supports documentation by objectifying the measurements and increasing transparency
* Improvement of the writing competence of the primary target group
* Increase of motivation and adherence to therapy sessions

The following research questions serve to evaluate the performance, as well as the functionality of the overall system, and its acceptance and effects. Sub-questions are listed as examples using bullet points.

Technical performance and functionality of the system

1.1: What technical performance does the system achieve in the everyday life of the target groups?

Usability of the system

2.1 How is usability described? What barriers exist in the real use of the individual components?

Acceptance of the system

3.1 Based on the UTAUT2 model, how are acceptance factors of the system evaluated by the target groups?

Effects of the system

4.1: What are the intended and unintended effects of the system for children, occupational therapists and legal guardians?

* Does the biofeedback improve the child's pressure behavior (finger pressure or mine pressure)?
* Does the system positively influence the motivation and adherence of the children?
* Does the system improve the child's graphic motor skills or handwriting based on the SEMS?
* Does the system increase the efficiency of the therapy (e.g. by eliminating documentation tasks)?

Study Design

The study uses a mixed-methods design. To quantitatively assess effectiveness, the study uses a Single Case Experimental Design (SCED) (Krasny-Pacini & Evans, 2018). Compared to the number of participants in existing SCED studies, the group size of n=15 (children only) is sufficiently large.

The number of participants for the qualitative data collection is n=15 per target group (occupational therapists, children, and legal guardians). Due to the deliberately narrow scope of the inclusion criteria, a certain homogeneity of the individual participant groups, based on their experiences, can be assumed (Guest, Bunce & Johnson, 2006). Romney, Batchelder, and Weller (1986) emphasize that small samples can be sufficient to provide complete and accurate information in a given context as long as participants have some level of expertise in the area of inquiry. Furthermore, Guest, Bunce, and Johnson (2006) suggest that if the homogeneity of the groups being studied is present, a participant count of 12 can generate sufficient saturation.

Methods

The research questions already mentioned are used for evaluation. The following overview of methods compares the evaluation factors used with the respective methods. Furthermore, it illustrates which users contribute to the evaluation of which questions in which study phase.

Evaluation of performance, usability and acceptance in the field Performance, usability and acceptance in the field will be determined on one hand via usage diaries and final interviews, and on the other hand via questionnaires based on the USE questionnaire and the UTAUT2.

i. Children (primary target group) contribute to the topic-specific knowledge gain

* by completing two short child-friendly questionnaires
* as well as by participating in the final interview.

ii. Occupational therapists (secondary target group) contribute to the topic-specific knowledge gain by

* documenting any errors and abnormalities in the use of the SensoGrip-System in therapy,
* filling out the USE and UTAUT2-based questionnaire after the intervention phase
* participating in the final interview

iii. Legal guardians (tertiary target group) contribute by

* completing the pre-questionnaire and
* completing the post-questionnaire (if the SensoGrip-Pen was given to them at home).

Evaluation of effects in the field

A Single Case Experimental Design (SCED) was chosen, to investigate the effectiveness of the intervention with the SensoGrip-System intrapersonally or on a small number of individuals, was chosen. In this approach, data from participating children will be studied prospectively and intensively. The outcome is measured repeatedly and multiple times throughout all phases of the study (Krasny-Pacini & Evans, 2018). The repeated measurements make it possible to detect effects in individuals or in groups of individuals; thus, the subjects represent their own control group. The design is especially suitable when studies are conducted in natural practice settings (Romeiser et al., 2017).

The exact structure of the design used in this study is as follows:

The study is divided into two phases (A/B):

Phase A - Baseline measurements

• Time point 0: Children are included in the study if the inclusion and exclusion criteria have been screened by the occupational therapist and the Informed Consent has been signed by a legal guardian and the participating child or the child has given oral informed consent. In addition to this, the pre-questionnaire of the legal guardian and the data sheet of the child will be filled in at time point 0.

• Time point 1: In the first regular therapy session after inclusion, the start of the baseline survey takes place. Preceding the start of regular therapy, the assessment instrument for the systematic evaluation of motor writing disorders (SEMS) is administered to children from 2nd grade on and a sheet of standard forms to children in 1st grade. Baseline measurement is recorded with SensoGrip using no feedback. This is followed by the regular therapy session. In the last five minutes of therapy, a standard sentence (from SEMS) or the standard forms are copied with the SensoGrip without feedback, but with data recording. To get used to the pen, drawing is done with the pen before writing down the test sentence.

• Timepoint 2: At the beginning and at the end of the session the chosen standard set is written down once with SensoGrip without feedback activated. To get used to the pen, the test set is drawn with the pen before writing it down.

Occupational therapists determine the first possible threshold values from the baseline data, which are used in the next sessions.

Phase B - Intervention phase

• Time point 3 - 7: From the third therapy session on, the child receives an explanation how SensoGrip works and is given feedback via a luminous ring at the tip of the SensoGrip-pen. Therapists now also receive the child's writing evaluation. At least 10 minutes per session should be spent working with SensoGrip. Possible sample exercises are provided, nevertheless therapists can use SensoGrip for other case-specific exercises aimed at improving pressure. Therapists document which exercises have been done and which adjustments have been made or tried. At the end of each session, the standard set is copied twice - once with and once without feedback. The order changes each time to minimize possible bias due to the order and thus habituation to writing with the pen. Data is recorded in both forms. Chosen settings are noted and selected as the therapist deems appropriate.

Optionally, the child can take the SensoGrip home starting from the fourth session and use it freely in everyday life, while the tablet remains with the therapist.

• Time point 8: In the last session SEMS or the standard forms are reevaluated. Writing is performed with the SensoGrip without feedback, but with data recording.

After completion of the intervention, an interview will be conducted individually with the participating children and the participating occupational therapists according to the interview guideline.

Parents or legal guardians will only receive a second questionnaire after the end of phase B if the SensoGrip pen was taken home and used there.

Intended outcomes of the study

The intended outcomes are focused on the following domains:

* Improve the writing skills of the primary target group The SensoGrip-System provides a feedback opportunity for training fine motor skills, visuomotor skills and kinesthesia. It is intended to support holding the pen with appropriate pressure and to write loosely / without tensing up. The system aims to increase motivation and adherence to therapy sessions through direct feedback. Subsequently, if therapy is successful, patients' performance at school could also be improved. Self-esteem of patients also plays an important role, which could be positively influenced by the improvement of writing competence.
* Improvement of the therapeutic possibilities Depending on the patient's needs, a new tool is available that has the potential to increase motivation and adherence to graphomotor exercises. Furthermore, after successful completion of the project, a tool enabling standardized diagnostics of graphomotor difficulties and visualization of therapeutic progress will be available. Through these improved possibilities of monitoring therapeutic processes, treatment progress can be made more measurable and thus also reported to health insurance companies by means of concrete figures.

ELIGIBILITY:
Inclusion Criteria:

Children

Participating children are between the ages of 5-10 years, and - if already in occupational therapy - have at least six more therapy sessions planned. Participating children must be motivated to participate in the study and have difficulties in graphomotor skills, of which at least two of the following criteria must apply:

* The child complains of pain when writing/drawing.
* The child's knuckles turn white due to high grip pressure when writing.
* The distal interphalangeal joint of the index and or middle finger is severely hyperextended when writing / drawing
* The writing imprints on the next page when writing / drawing
* The child has to take regular breaks when writing / drawing in order to relax the hand.
* The child's hand slides to the tip of the pencil when writing / drawing because the pencil is held too loosely
* The child's writing/drawing is difficult to see because too little pressure is being applied
* The pen slips out of the child's hand when writing / drawing
* The child cannot guide the pencil sufficiently because it is held too loosely
* The child frequently breaks the pencil lead while writing or drawing or pushes a felt-tip pen lead into the pencil.
* Grip pressure or pressure on the paper varies greatly during writing / drawing

Other than the graphomotor problems, participating children must have the following cognitive abilities to participate in the study:

* Sufficient language and task comprehension to follow instructions
* Ability to follow simple verbal instructions
* Maintenance of attention for 10 minutes during graphomotor activities at the table

In addition, the following motor skills must be present to hold the pencil:

* No stiffened joints in the finger and hand area (sufficient gripping function and finger mobility), so that it is possible to both hold objects in the hand and move them while holding them in the hand.
* No excessive or insufficient muscle tension at rest (hyper-/hypotonia) in the upper extremities or writing hand, so that it is possible to hold a pen in the hand.

Additionally, participating children must confirm their consent to participate in the study in writing via a child-friendly Informed Consent (IC) form. Furthermore, a parent/guardian must confirm the child's participation in the parent/guardian IC by signature in each case.

Occupational Therapists

Participating occupational therapists possess at least two years of professional experience in the occupational therapy assessment and treatment of children, in which context participants also treat children with graphomotor problems in an activity-based manner. Furthermore, the participating occupational therapists have at least average technical affinity (handling of a normal tablet is possible). Occupational therapists will only be involved if the IC has been completed and signed.

Legal Guardians

Legal guardians are included if the IC has been filled out completely, signed and if participants have at least average technical affinity (necessary in case of "home use" of the SensoGrip pen by the child).

Exclusion Criteria:

Children

Children will be excluded from participating in the study if there is a concurrent participation in another study related to graphomotor skills, their age is inappropriate, the adequate development of motor and cognitive skills is not present, or if there are significant problems in the area of psychosocial skills such as critical thinking skills, emotion regulation, or frustration tolerance.

Occupational Therapists

Occupational therapists will not be recruited for the study if their work with children is exclusively focused on the gross motor area, therapists are specialized in other areas and do not have sufficient professional experience. Further exclusion criteria are the rejection of technical tools in therapy and serious uncertainties or fears in the use of technologies.

Legal Guardians

Legal guardians are excluded if participants generally reject the use of technical devices or have serious insecurities or fears regarding the use of the technology.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Sum of the finger-pressure readings on the pen's surface in milligram via a written standardized sentence | 6-8 weeks
Sum of the tip-pressure readings of the pen against the paper in milligram via a written standardized sentence | 6-8 weeks

SECONDARY OUTCOMES:
Usability of the SensoGrip-System | 6-8 weeks
  Data regarding the usability of the SensoGrip-System is collected via usage diaries, interviews the USE-based and the post questionnaire
Acceptance of the SensoGrip-System | 6-8 weeks
  Data regarding the acceptance of the SensoGrip-System is collected via the UTAUT2-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Franz Werner, Dr., Study Director — FH Campus Wien - University of Applied Life Sciences
Locations (1):
- FH Campus Wien - University of Applied Life Sciences Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart SR. Development of written language proficiency: methods for teaching text structure. In: Simon CS, editor. Communication Skills and Classroom Success. Eau Claire, WI: Thinking Publications. 1992; 419-432
- [Background] Sassoon R. Handwriting: A New Perspective. Cheltenham, UK: Stanley Thornes. 1990
- [Background] Kruse, O. Schlüsselkompetenz Schreiben: Konzepte, Methoden, Projekte für Schreibberatung und Schreibdidaktik an der Hochschule. Hochschulwesen - Wissenschaft und Praxis. Luchterhand. 1999
- [Background] Diaz Meyer, M., Marquardt, C. & Klimen, A. (2017). Die Rolle der Schreibmotorik beim Schreibenlernen. Eltern und Lehrer beunruhigt. Ergotherapie und Rehabilitation, 56 (10), 18-21.
- [Background] Karlsdottir R, Stefansson T. Problems in developing functional handwriting. Percept Mot Skills. 2002 Apr;94(2):623-62. doi: 10.2466/pms.2002.94.2.623. PMID 12027360
- [Background] Hoy MM, Egan MY, Feder KP. A systematic review of interventions to improve handwriting. Can J Occup Ther. 2011 Feb;78(1):13-25. doi: 10.2182/cjot.2011.78.1.3. PMID 21395194
- [Background] Schneck, C. M. & Case-Smith, J. Prewriting and Handwriting Skills. In J. Case-Smith & J. C. O'Brien (Hrsg.), Occupational therapy for children 2014; 498-524.
- [Background] Dolezal, D. & Schönthaler, E. Ergotherapie bei Kindern und Jugendlichen mit umschriebener Entwicklungsstörung motorischer Funktionen in Österreich - eine Umfrage. Schulz-Kirchner Verlag. 2018; https://doi.org/10.2443/skv-s-2018-54020180402
- [Background] Blank R., Vinçon S. Deutsch-österreichisch-schweizerische (DACH) Versorgungsleitlinie zu Definition, Diagnostik,Behandlung und psychosozialen Aspekten bei Umschriebenen Entwicklungsstörungen motorischer Funktionen (UEMF), Langfassung. Arbeitsgemeinschaft der Wissenschaftlichen Medizinischen Fachgesellschaften (AWMFonline);2020)
- [Background] Gaines R, Missiuna C, Egan M, McLean J. Interprofessional care in the management of a chronic childhood condition: Developmental Coordination Disorder. J Interprof Care. 2008 Oct;22(5):552-5. doi: 10.1080/13561820802039037. No abstract available. PMID 24567970
- [Background] Blank R, Smits-Engelsman B, Polatajko H, Wilson P; European Academy for Childhood Disability. European Academy for Childhood Disability (EACD): recommendations on the definition, diagnosis and intervention of developmental coordination disorder (long version). Dev Med Child Neurol. 2012 Jan;54(1):54-93. doi: 10.1111/j.1469-8749.2011.04171.x. No abstract available. PMID 22171930
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders. American Psychiatric Association. 2013; https://doi.org/10.1176/appi.books.9780890425596
- [Background] Maeland AF. Handwriting and perceptual-motor skills in clumsy, dysgraphic, and 'normal' children. Percept Mot Skills. 1992 Dec;75(3 Pt 2):1207-17. doi: 10.2466/pms.1992.75.3f.1207. PMID 1484789
- [Background] Lin YC, Chao YL, Wu SK, Lin HH, Hsu CH, Hsu HM, Kuo LC. Comprehension of handwriting development: Pen-grip kinetics in handwriting tasks and its relation to fine motor skills among school-age children. Aust Occup Ther J. 2017 Oct;64(5):369-380. doi: 10.1111/1440-1630.12393. Epub 2017 May 16. PMID 28512858
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Guest, G., Bunce, A., & Johnson, L. How many interviews are enough? An experiment with data saturation and variability. Field methods. 2006; 18(1), 59-82.
- [Background] Romney, A., W. Batchelder, and S. Weller. Culture as consensus: A theory of culture and informant accuracy. American Anthropologist. 1986; 88:313-38.
- [Background] Romeiser-Logan L, Slaughter R, Hickman R. Single-subject research designs in pediatric rehabilitation: a valuable step towards knowledge translation. Dev Med Child Neurol. 2017 Jun;59(6):574-580. doi: 10.1111/dmcn.13405. Epub 2017 Feb 22. PMID 28224606